CLINICAL TRIAL: NCT05467800
Title: A Phase 2 Study of Canakinumab in Patients With Myelofibrosis Myeloproliferative Neoplasms Research Consortium [MPN-RC 122]
Brief Title: Study of Canakinumab in Patients With Myelofibrosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: John Mascarenhas (Other)
Responsible Party: Sponsor-Investigator, John Mascarenhas, Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 22-0543; MPN-RC 122 (Other: The Myeloproliferative Neoplasms Research Consortium (MPN-RC))
Record Dates: First submitted 2022-07-18; First posted 2022-07-21 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Primary Myelofibrosis; Post-essential Thrombocythemia Myelofibrosis; ET-MF; Post-polycythemia Vera Related Myelofibrosis; PV-MF
MeSH Terms: conditions — Primary Myelofibrosis | interventions — canakinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Canakinumab (Experimental): Canakinumab will be given by subcutaneous injection (SC) injection at a starting dose of 200 mg (one 150 mg/mL syringe and one 50 mg/0.5 mL syringe) every 3 weeks.
  Interventions: Drug: Canakinumab

INTERVENTIONS:
Drug: Canakinumab — Canakinumab administered as a subcutaneous injection on day 1 of a 21 day cycle for a core study period of 8 cycles.

SUMMARY:
This is an open label, multicenter, phase 2 trial of Canakinumab in patients with primary myelofibrosis (PMF), post essential thrombocythemia/polycythemia vera related MF (Post ET/PV MF). Eligible patients will receive Canakinumab administered as a subcutaneous injection on day 1 of a 21 day cycle for a core study period of 8 cycles. Canakinumab will be given by subcutaneous injection (SC) injection at a starting dose of 200 mg (one 150 mg/mL syringe and one 50 mg/0.5 mL syringe) every 3 weeks. The interim analysis will be performed when the number of enrolled patients reaches 10. If no responses OR 4 or more patients have unacceptable toxicity, the study will not proceed to the second stage. If the total number of patients reaches the maximum sample size of 26, the treatment is deemed acceptable if the number of responses in the efficacy endpoint are greater than 3, and the number of toxicities are less than 7.

ELIGIBILITY:
Inclusion Criteria

The following are required for inclusion in the study:

Parts 1 and 2:

1. Participants must voluntarily sign informed consent form (ICF) and be willing and able to adhere to the study visit schedule and all protocol requirements.
2. Participants must be ≥ 18 years of age at the time of signing the ICF.
3. Participants must have a pathologically confirmed diagnosis of PMF as per the World Health Organization (WHO) diagnostic criteria46 or post-ET MF or post-PV MF according to IWG-MRT criteria.47
4. Participants must have at least one of the following:

   1. Hemoglobin < 10 g/dL
   2. Transfusion-dependency (at least 6 units of packed red blood cells (PRBC) in the 12 weeks prior to study enrollment, for a hemoglobin < 8.5 g/dL, in the absence of bleeding or treatment-induced anemia with the most recent transfusion having occurred in the 28 days prior to study enrollment)
   3. Splenomegaly palpated ≥ 5 cm below the left costal margin (LCM) or spleen volume ≥ 450 cc
   4. MFSAF v4.0 TSS ≥ 10
5. A bone marrow biopsy must be performed within the 30-day screening period; however, a bone marrow biopsy obtained within 90 days of signing ICF without intervening treatments and approved by the study chair may suffice.
6. Participants must have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2.
7. Life expectancy of at least 6 months.
8. Recovery to ≤ Grade 1 or baseline of any toxicities due to prior systemic treatments excluding alopecia.
9. Women of childbearing potential (WCBP) must have a negative urine or serum pregnancy test within 28 days of starting the study drug. Men and women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence, tubal ligation, vasectomy) prior to Cycle 1 Day 1 and for 130 days after stopping study treatment. Vasectomy must be performed a minimum of 3 months before study start.
10. Must have adequate organ function as demonstrated by the following:

    1. ALT/AST ≤ 3.0 x ULN, or ≤ 4 x ULN (unless if upon judgment of the treating physician, it is believed to be due to EMH related to MF);
    2. Direct bilirubin ≤ 1.5 x ULN or ≤ 2.0 x ULN (unless if upon judgment of the treating physician, it is believed to be due to EMH related to MF or documented Gilbert's syndrome);
    3. Serum creatinine ≤ 2.0 mg/dL;
    4. Platelet count ≥ 25 x 109/L (participant must not have had platelet transfusion in the 14 days prior to signing ICF);
    5. ANC ≥ 1000/µL
11. Participant must be willing to receive red blood cell and/or platelet transfusions if indicated.
12. Bone marrow and peripheral blood blast count < 10%.

    Part 1 Only:
13. At least two weeks must have elapsed between the last dose of any MF-directed drug treatments (including investigational therapies and excluding hydroxyurea) and study enrollment.
14. Not eligible for available, approved JAKi therapy due to a platelet count of < 50 x 109/L or previously treated and lack/loss of response per investigator discretion.

    Part 2 Only:
15. Current treatment with a JAKi (inclusive of ruxolitinib, fedratinib, momelotinib, or pacritinib) for at least 16 weeks and on a stable or decreased dose for at least 12 weeks prior to study enrollment.

Exclusion Criteria

Any of the following is a criterion for exclusion from the study:

1. Prior malignancy active within the previous ≤ 1 year except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast.
2. Any of the following cardiac abnormalities

   1. Uncontrolled, symptomatic congestive heart failure as designated by the treating physician
   2. Myocardial infarction ≤ 6 months prior to enrollment
   3. Unstable angina pectoris designated by treating physician
   4. Serious uncontrolled cardiac arrhythmia as designated by treating physician
   5. Uncontrolled hypertension as designated by treating physician
3. Known history of human immunodeficiency virus (HIV) (no laboratory testing is required), or active infection with hepatitis B or Hepatitis C.
4. Active TB infection or documented, untreated latent TB infection (all participants should undergo TB risk evaluation prior to enrollment with TB screening performed as per local guidelines.)
5. Active, uncontrolled infection at the time of enrollment, except in cases of localized infections that are unlikely to lead to a systemic infection such as onychomycoses or dental caries.

   a. Participants with a new fever (T>38.0o C) or respiratory symptoms are required to undergo laboratory screening for COVID-19.
6. Have undergone prior allo-HSCT for treatment of any hematological disorder or prior solid organ transplant
7. Any serious or uncontrolled psychiatric or medical disorder that, in the opinion of the investigator, may increase the risk associated with the study participation or study drug administration, impair the ability of the participants to receive protocol therapy, or interfere with the interpretation of study results.
8. Women who are pregnant or breastfeeding.
9. Participants undergoing concurrent treatment with agents targeting TNF-α or IL-1 within 28 days of study enrollment.
10. Participants who have received a live vaccination within 90 days before study drug administration (participants should not be treated with live-virus vaccine while undergoing therapy and 130 days after Canakinumab discontinuation).
11. Participants with a condition requiring systemic treatment with corticosteroids within 14 days of study drug administration (i.e. prednisone at doses of > 10 mg). Inhaled or topical steroids and adrenal/pituitary replacement doses ≤ 10mg daily of prednisone or equivalent are permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2022-08-02 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of participant with response based on IWG-MRT criteria | 24 weeks
  Efficacy of Canakinumab as measured by number of participant with response based on the International Working Group for Myelofibrosis Research and Treatment (IWG-MRT) criteria. A response is considered any one of the following: complete response, partial response, or clinical improvement (inclusive of anemia response, spleen response, or symptom response).

SECONDARY OUTCOMES:
Number of Adverse Events | 24 weeks
  The safety and tolerability of Canakinumab as measured by the adverse event profile of Common Terminology Criteria for Adverse Events version 5.0
Response using IWG-MRT | 12 weeks
  To assess the efficacy of Canakinumab as determined by response assessment using IWG/ELN criteria. Participant's response will be categorized as negative, stable, or positive.
Response using IWG-MRT | 24 weeks
  To assess the efficacy of Canakinumab as determined by response assessment using IWG/ELN. Participant's response will be categorized as negative, stable, or positive.
Number of participants with clinical improvement | 12 weeks
  Clinical improvement (CI) is defined by IWG-MRT criteria. Participants meet CI if meet any of the following:
  Anemia (Patients will meet IWG-MRT criteria for clinical improvement if their hemoglobin increase by 2g/dl from baseline and/or become transfusion independent.)
  Splenomegaly (Patients will meet IWG-MRT criteria for clinical improvement if their spleen decreases by ≥30% from baseline volume.)
  Disease-related symptoms (Patients will meet IWG-MRT criteria for clinical improvement if their MPN-SAF symptom score decreases by ≥50% from baseline)
Number of participants with clinical improvement | 24 weeks
  Clinical improvement (CI) is defined by IWG-MRT criteria. Participants meet CI if meet any of the following:
  Anemia (Patients will meet IWG-MRT criteria for clinical improvement if their hemoglobin increase by 2g/dl from baseline and/or become transfusion independent.)
  Splenomegaly (Patients will meet IWG-MRT criteria for clinical improvement if their spleen decreases by ≥30% from baseline volume.)
  Disease-related symptoms (Patients will meet IWG-MRT criteria for clinical improvement if their MPN-SAF symptom score decreases by ≥50% from baseline)
Change in Spleen Volume | 12 weeks
  Change in Spleen Volume as compared to baseline
Change in Spleen Volume | 24 weeks
  Change in Spleen Volume as compared to baseline
Overall Survival (OS) | 24 weeks
  OS is defined as the time from the first dose of study treatment to the date of death (whatever the cause).
Progression free survival (PFS) | 12 weeks
  PFS is defined as the duration of time from start of treatment to the first occurrence of disease progression or death on study from any cause, whichever occurs earlier.
Progression free survival (PFS) | 24 weeks
  PFS is defined as the duration of time from start of treatment to the first occurrence of disease progression or death on study from any cause, whichever occurs earlier.

CONTACTS AND LOCATIONS:
Overall Officials: John Mascarenhas, MD, Study Chair — MOUNT SINAI HOSPITAL
Locations (8):
- United States (8):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Cedars-Sinai Medical Center, Samuel Oschin Comprehensive Cancer Institute, Los Angeles, California
  - Moffitt Cancer Center, Tampa, Florida
  - The University of Kansas Cancer Center-Westwood, Westwood, Kansas
  - Ruttenberg Treatment Center, New York, New York
  - Atrium Health Levine Cancer Institute, Charlotte, North Carolina
  - Wake Forest Baptist Health Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No